CLINICAL TRIAL: NCT00324896
Title: Treatment of Insomnia in Patients With Parkinson's Disease: A Multi-site, Placebo-controlled Study of Eszopiclone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5581
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson's Disease; Insomnia
Keywords: Parkinson's; insomnia; drug; eszopiclone; placebo
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- eszopiclone (Experimental): eszopiclone. Those under 65yo received 3mg of eszoplicone ( or randomized to matching placebo)and those 65yo or older received 2mg of eszoplicone ( or randomized to matching placebo)taken each night at bedtime
  Interventions: Drug: eszopiclone
- placebo (Placebo Comparator): Those randomly assigned to matching placebo, took their dose each night at bedtime
  Interventions: Other: placebo

INTERVENTIONS:
Drug: eszopiclone — eszopiclone
  Other Names: Lunesta 2 - 3 mg q HS
  Arms: eszopiclone
Other: placebo — matching placebo administered at night
  Arms: placebo

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease in the US, affecting nearly 1 million Americans. Up to 82% of community dwelling individuals with PD complain of sleep disturbances, typically sleep fragmentation. Despite the high prevalence of sleep problems and their impact on the life of these individuals, there has been, until recently, little research focus on the problem. This will be a multi-site, double blind, placebo-controlled, two arm, parallel group, fixed-dose trial which will last 6 weeks. Seventy patients at four sites (30 at the PI's site and a total of 40 patients at three external sites) will be equally randomized to eszopiclone or placebo. The primary hypothesis is that eszopiclone will be superior to placebo for the treatment of insomnia in patients with Parkinson's disease

DETAILED DESCRIPTION:
Introduction and Rationale Parkinson's disease (PD) is the second most common neurodegenerative disease in the US, affecting nearly 1 million Americans. Up to 82% of community dwelling individuals with PD complain of sleep disturbances, typically sleep fragmentation. This difficulty with sleep maintenance is accompanied by a decrease in total sleep time and an increase in the number of awakenings and wakefulness after sleep. The interactions between PD and sleep are complicated and many PD patients with insomnia have concomitant sleep disorders such as REM Sleep Behavior Disorder (RBD), Periodic Limb Movements of Sleep (PLMS) and Sleep Disordered Breathing (SDB). Nonetheless, the majority of patients appear to have insomnia that is an integral symptom of PD rather than being related to specific sleep disorders. Sleep difficulties in patients with PD are independent and important predictors of poor quality of life. In addition, sleep disturbances contribute to excessive daytime sleepiness (EDS) and poor daytime functioning as well as patients' reduced enthusiasm for daily events and impairment in the quality of life of their spousal caregivers7. There are, therefore, a variety of reasons for us to address sleep problems in patients with PD.

Despite the high prevalence of sleep problems and their impact on the life of these individuals, there has been, until recently, little research focus on the problem. While researchers have now begun to describe the phenomenology and epidemiology of sleep in PD, there have few treatment studies from which the clinical community can derive guidance. Despite this lack of evidenced-based clinical guidance, community surveys indicate that up to 40% of patients with PD are taking sleeping pills.3 Data published in 1999 indicate that the two most commonly used hypnotics in general practice were trazodone and zolpidem. More recent data continue to show that trazodone is prescribed even more frequently than zolpidem. We have recently completed a survey of 50 Parkinson's disease experts and found that the most commonly used hypnotics were zolpidem and trazodone. Of note is also that these experts estimated that 40% of their patients with PD were using sleep medications.

We have then the following clinical problem in the treatment of patients with PD. Insomnia is very common and is strongly associated with a variety of adverse outcomes but there are no controlled data that can guide the approach to the treatment of these individuals. Nevertheless, clinicians appear to be using a number of hypnotics, principally zolpidem and trazodone, neither of which have been evaluated in PD or for long term use.

Objectives

To test the safety and efficacy of eszopiclone for the treatment of insomnia in patients with Parkinson's disease

Hypothesis

Eszopiclone will result in significantly greater improvement than placebo in patient reported total sleep time (diaries) in patients with PD in an six week trial.

Study Design and Duration

This will be a multi-site, double blind, placebo-controlled, two arm, parallel group, fixed-dose trial which will last 6 weeks. Seventy patients at four sites (30 at the PI's site and a total of 40 patients at three external sites) will be equally randomized to eszopiclone or placebo.

Preliminary screening will be conducted by telephone. Inclusion and exclusion criteria are listed below. Those individuals appearing appropriate will be scheduled for an in-person screening visit and will sign informed consent. At the screening visit, a detailed sleep, medical and psychiatric history, and a variety of background demographic forms (See Schedule of Events - Appendix A) will be completed.

Subjects meeting all entrance criteria will be scheduled for a polysomnogram at the end of a two-week baseline period during which they will keep sleep-wake diaries. Those who meet criteria for insomnia receive overnight polysomnographic evaluations to screen for primary sleep disorders of REM Sleep Behavior Disorder (RBD), Periodic Limb Movements of Sleep (PLMS), and Sleep Disordered Breathing (SBD). To minimize cost, we plan to obtain one or two nights of baseline PSG evaluation, depending on the amount of total sleep time observed on the first night of recording. Patients who show 4 hours or more of total sleep, including at least 30 min total of REM sleep, will receive only one night of PSG evaluation. These values were selected as the minimum necessary amount of sleep for evaluating concomitant sleep disorders. Patients who do not meet these criteria on the first night, or whose results are equivocal, will receive a second night of baseline evaluation. The exclusion criteria will apply to the either night. If there is not sufficient sleep on either night the patient will be excluded.

Polysomnographic evaluation will be conducted using standard nocturnal polysomnographic procedures. This consists of 2 monopolar electroencephalographic (EEG) leads (C3-A2 and O1-A2), 2 monopolar electro-oculograms (EOG), bipolar submental (chin) and right and left tibialis (leg) electromyograms (EMG), and electrocardiogram (ECG). Respiratory airflow will be monitored through the use of a thermocouple (Pro-Tech Services, Inc.), placed at the nose and mouth. Respiratory effort will be measured by plethysmography using piezoelectric sensors (Pro-Tech Services, Inc.) Snoring will be recorded through the use of a snoring sensor (Pro-Tech Services, Inc.). Arterial oxygen saturation will be measured with a finger probe and pulse oximeter (Nonin). All subjects will be videotaped during the PSG evaluation to provide positional and behavioral information regarding their sleep episode. All sleep parameters will be collected simultaneously by a computerized acquisition system (REMbrandt, Medcare Diagnostics). Sleep will be scored in 30-second epochs according to the standard criteria of Rechtschaffen and Kales.

Those meeting entrance criteria will then be equally randomly assigned to receive eszopiclone or placebo treatment for 6 weeks. Both groups will receive equal-appearing pills to be taken each night. The dosing in the trial will be fixed and stratified by age: those under 65 will receive 3 mg of eszopiclone or matching placebo at night; those 65 or older will receive 2 mgs of eszopiclone or placebo at night.

Patients will have visits at screen, an interim phone contact to review the sleep diaries, PSG, baseline and weeks 2, 4, and 6, at which medication will be monitored and pill intake, therapeutic response and adverse events will be reviewed. The procedures done at each visit are listed in Appendix A. All groups will record sleep-wake diaries during the 2 week screening phase and for the first six weeks of the study.

Patients will be asked but not be required to provide a care giver who will complete questionnaires at the screen visit and week 6 visit.

Patients who terminate prematurely or who continue in the trial till the end will stop medication and continue to record diaries for one week at which time they will return for the final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease by research criteria. Research criteria for PD include, (1) the presence of at least 2 of the following signs: resting tremor, cogwheel rigidity, bradykinesia, or postural reflex impairment, at least 1 of which must be either resting tremor or bradykinesia, (2) no other cause of parkinsonism, (3) no signs of more extensive neurodegeneration indicating atypical parkinsonism, and (4) a clear-cut response to levodopa or dopamine agonist.
2. Sleep maintenance insomnia (at least 3 of 7 nights of at least 2 awakenings nightly, or a total sleep time of < 6.5 hours) or sleep latency insomnia (at least 3 of 7 nights of sleep latency > 30 minutes), as well as clinically significant daytime distress or impairment during the 2 week self assessment prior to baseline.
3. Patients aged 35-85 years.
4. Patients must have completed at least the 9th grade and be fluent in English.
5. If a female of child bearing potential, the patient must be non-pregnant and either post-menopausal or using an approved birth control method. Patients must have a negative urine pregnancy test at the screen visit.
6. Antidepressants will be allowed if the patient has been on a stable dose for at least one month.
7. Benzodiazepines will be allowed if taken during the day prior to 6pm and it is not taken as a sleep aid.
8. Other medications with CNS activity that the patient is on at screening, e.g., dopaminergic drugs, B-blockers, etc, will be kept constant throughout the acute phase.

   -

Exclusion Criteria:

1. Evidence on PSG and symptoms or complaints (as defined below) of, significant sleep disordered breathing (central or obstructive apnea), periodic limb movement disorder (PLMD), or REM sleep behavior disorder (RBD).
2. Significant sleep disordered breathing will be defined as an AHI > 15 events/hr of sleep and/or significant hypoxemia on screening PSG; significant PLMD will be defined as a PLM index > 25 events/hr of sleep on screening PSG; RBD will be defined based on presence of both clinical symptomatology (demonstrated injury to self or others during sleep) as well as PSG criteria (intermittent loss of REM atonia).
3. No significant dementia. Significant dementia is operationalized as a score of less than 26 on the Mini-Mental State Examination (MMSE).
4. Insomnia is not primarily due to serious depression or anxiety in the opinion of the investigator.
5. Any current (within three months) diagnosis of alcohol or substance abuse/dependence (with the exception of nicotine dependence).
6. Currently on psychotropic medications, other than antidepressants or benzodiazepines. If the patient is on other psychotropics, and can be safely removed from these medications at the time of initial screening, there will be a washout period prior to entering the study.
7. Sleep medication that the patient is on during screening will be tapered prior to randomization.
8. Any unstable medical disorder that would interfere with the study.
9. Patients with a known history of non-response or lack of toleration to adequate doses of zolpidem or trazodone.
10. Patients currently receiving CBT for insomnia.
11. Patients who are unable to be maintained on their current dose of PD medications throughout the trial.

    -

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Menza, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (4):
- United States (4):
  - Fusion Sleep Center, Suwanee, Georgia
  - The New Jersey Neuroscience Institute, Edison, New Jersey
  - UMDNJ Robert Wood Johnson Medical School, Piscataway, New Jersey
  - University of Pennsylvania Medical School, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Menza M, Dobkin RD, Marin H, Gara M, Bienfait K, Dicke A, Comella CL, Cantor C, Hyer L. Treatment of insomnia in Parkinson's disease: a controlled trial of eszopiclone and placebo. Mov Disord. 2010 Aug 15;25(11):1708-14. doi: 10.1002/mds.23168. PMID 20589875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 2006 and 2009, from the RWJMS movement disorder clinic and advertising to local support groups.
Pre-assignment Details: Patients who met inclusion and exclusion criteria were enrolled.
Groups:
- Eszopiclone: eszopiclone. Those under 65yo received 3mg of eszoplicone (or randomized to matching placebo)and those 65yo or older received 2mg of eszoplicone (or randomized to matching placebo)taken each night at bedtime
  eszopiclone : eszopiclone
Period: Overall Study
Arm/Group | Eszopiclone | Placebo
Started | 15 | 15
Completed | 12 | 7
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 4 | 5 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.9) | 53.1 (10.5) | 56.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: TST
Description: Total sleep time in hours
Time Frame: 6 weeks
Population: intent to treat approach
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 15 | 15
hours | 5.7 (1.16) | 6.0 (1.16)

2. Secondary Outcome: WASO
Description: Wake after sleep onset in minutes
Time Frame: 6 weeks
Population: intent to treat
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 15 | 15
minutes | 17 (50) | 46 (45)

ADVERSE EVENTS:
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone (N=15) | Placebo (N=15)
sedation (Nervous system disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) — One patient experienced both dizziness and sedation
daytime fatigue (Nervous system disorders) | 0 (0) | 3 (3)
increase Parkinson's related rigidity (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was only a 6-week trial with small group of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No